CLINICAL TRIAL: NCT06151288
Title: A Phase 1/2, Randomized, Observer-Blind, Dose-Finding, Active-Controlled, Parallel-Group, Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of a 31-Valent Pneumococcal Conjugate Vaccine (VAX-31) in Healthy Adults Aged 50 Years and Older
Brief Title: Safety, Tolerability, and Immunogenicity Study of a 31-Valent Pneumococcal Conjugate Vaccine (VAX-31) in Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vaxcyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAX31-101
Record Dates: First submitted 2023-11-10; First posted 2023-11-30 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Participants received a single low dose of VAX-31 administered as an intramuscular injection at Day 1.
  1.1 mcg for all serotypes with the exception of serotypes 1, 5, and 22F which is 1.65 mcg.
  Interventions: Biological: 31 valent pneumococcal conjugate vaccine
- Group 2 (Experimental): Participants received a single mid dose of VAX-31 administered as an intramuscular injection at Day 1.
  2.2 mcg for all serotypes with the exception of serotypes 1, 5, and 22F which is 3.3 mcg.
  Interventions: Biological: 31 valent pneumococcal conjugate vaccine
- Group 3 (Experimental): Participants received a single high dose of VAX-31 administered as an intramuscular injection at Day 1.
  3.3 mcg for all serotypes with the exception of serotypes 1, 5, and 22F which is 4.4 mcg.
  Interventions: Biological: 31 valent pneumococcal conjugate vaccine
- Group 4 (Active Comparator): Participants received a single intramuscular injection of the standard dose of PCV20 at Day 1.
  Interventions: Biological: 20 valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 31 valent pneumococcal conjugate vaccine — 0.5 ml dose of VAX-31 was administered into the deltoid muscle at Day 1
  Arms: Group 1; Group 2; Group 3
Biological: 20 valent pneumococcal conjugate vaccine — 0.5 ml dose of PCV20 was administered into the deltoid muscle at Day 1
  Other Names: PCV20; Prevnar 20™
  Arms: Group 4

SUMMARY:
The objective of the study is to evaluate the safety, tolerability and immunogenicity of a single injection of VAX-31 at 3 dose levels compared to Prevnar 20™ (PCV20) in adults 50 to 64 years of age in Stage 1. Stage 2 will evaluate the safety, tolerability, and immunogenicity of a single injection of VAX-31 at 3 dose levels compared to PCV20 in adults aged 50 years and older.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 50 to 64 years (inclusive) for Stage 1, or 50 years and older (inclusive) for Stage 2 at the time of randomization into the study.
2. Able and willing to complete the informed consent process.
3. Available for clinical follow-up through the last study visit at 6 months after the study vaccination.
4. In good general health as determined by medical history, vital signs, physical examination, and clinical judgment of the Investigator.
5. Willing to have blood samples collected, stored indefinitely, and used for research purposes.
6. Able to provide proof of identity to the satisfaction of the study staff completing the enrollment process.
7. Women of childbearing potential, defined as premenopausal females capable of becoming pregnant, must have a negative urine pregnancy test immediately prior to randomization and agree to use acceptable contraception
8. Able to access and use a smartphone, tablet, computer, or other device connected to Wi-Fi or cellular network for completion of an electronic diary.

Exclusion Criteria:

1. Previous pneumococcal disease (either confirmed or self-reported).
2. Previous receipt of a licensed or investigational pneumococcal vaccine.
3. Receipt of any investigational study product within 30 days prior to enrollment into the study, currently participating in another interventional investigational study, or having plans to receive another investigational product(s) while on study.
4. Planned or actual administration of any licensed vaccine during the period starting 30 days before enrollment into the study through Month 1.
5. Physical examination indicating any clinically significant medical condition.
6. Body Temperature >38.0°C (>100.4°F) or acute illness within 3 days prior to study vaccination (subject may be rescheduled).
7. Previous or existing diagnosis of HIV, Hepatitis B, or Hepatitis C.
8. History of severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis.
9. Female who is pregnant, breastfeeding, or planning to become pregnant during study participation.
10. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) resulting in clinically significant bruising or bleeding difficulties with IM injections or blood draws.
11. Any other chronic or clinically significant medical condition that, in the opinion of the Investigator, would jeopardize the safety or rights of the subject or confound evaluation of the study vaccine.
12. Any medical, psychiatric, or social condition that in the judgment of the Investigator is a contraindication to protocol participation or impairs a subject's ability to give informed consent.
13. Received blood or blood product (including Immune Globulin IV) within 90 days prior to enrollment into the study.
14. Received systemic corticosteroids (except for inhaled, topical, intra-articular) for

    ≥14 consecutive days and has not completed treatment ≤30 days prior to enrollment into the study.
15. Receiving immunosuppressive therapy.
16. History of malignancy ≤5 years before enrollment, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Vaxcyte, Inc.
Locations (25):
- United States (25):
  - AMR Mobile, Mobile, Alabama
  - AMR Phoenix, Phoenix, Arizona
  - Research Centers of America, Hollywood, Florida
  - Health Awareness, Jupiter, Florida
  - Optimal Research, Melbourne, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - Healthcare Research Network II, LLC, Flossmoor, Illinois
  - Johnson County Clin-Trials, Lenexa, Kansas
  - DM Clinical Research - Detroit, Detroit, Michigan
  - Velocity Clinical Research Omaha, Omaha, Nebraska
  - WR-CRCN, Las Vegas, Nevada
  - Cenexel AMRI, Toms River, New Jersey
  - Rochester Clinical Research, Rochester, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Research, Cleveland, Cleveland, Ohio
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - Velocity Clinical Research, Warwick, Rhode Island
  - Coastal Carolina Research, North Charleston, South Carolina
  - AMR Knoxville, Knoxville, Tennessee
  - Benchmark Research, Fort Worth, Texas
  - Benchmark Research, San Angelo, Texas
  - CenExel JBR Clinical Research, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Health Research of Hampton Roads, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Vaxcyte is committed to providing access to anonymized data from the company's clinical trials for the purpose of legitimate scientific research. Requests for data may be addressed to datasharing@vaxcyte.com. Requests must be accompanied by a detailed analysis plan and will be reviewed for scientific validity. Data will be made available after initial product approval. Sharing of data may require execution of a data-sharing agreement.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be shared after deidentification and made available starting 6 months after initial product approval.
Access Criteria: Criteria will depend on the specific proposal received and may include qualification of the scientific researchers, potential contribution to the research field, scientific rigor of statistical and analytical methods, and other criteria appropriate for the proposal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was enrolled 08-Nov-2023 and last subject randomized/vaccinated was 10-Jan-2024. Study sites were medical clinics.
Pre-assignment Details: 1165 participants were screened. Of these, 150 failed screening, 98 did not meet eligibility criteria and 52 were excluded for other reasons. 13 participants were lost to follow-up and 11 withdrew from study.
Groups:
- VAX-31 Low Dose: Participants received a single low dose of VAX-31 administered as an intramuscular injection at Day 1.
  1.1 mcg for all serotypes with the exception of serotypes 1, 5, and 22F which is 1.65 mcg.
  31 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-31 will be administered into the deltoid muscle at Day 1
- VAX-31 Mid Dose: Participants received a single mid dose of VAX-31 administered as an intramuscular injection at Day 1.
  2.2 mcg for all serotypes with the exception of serotypes 1, 5, and 22F which is 3.3 mcg.
  31 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-31 will be administered into the deltoid muscle at Day 1
- VAX-31 High Dose: Participants received a single high dose of VAX-31 administered as an intramuscular injection at Day 1.
  3.3 mcg for all serotypes with the exception of serotypes 1, 5, and 22F which is 4.4 mcg.
  31 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-31 will be administered into the deltoid muscle at Day 1
- PCV20: Participants received a single intramuscular injection of the standard dose of PCV20 at Day 1.
  20 valent pneumococcal conjugate vaccine: 0.5 ml dose of PCV20 will be administered into the deltoid muscle at Day 1
Period: Overall Study
Arm/Group | VAX-31 Low Dose | VAX-31 Mid Dose | VAX-31 High Dose | PCV20
Started | 255 | 254 | 253 | 253
Completed | 247 | 247 | 248 | 249
Not Completed | 8 | 7 | 5 | 4
Not completed — Lost to Follow-up | 4 | 2 | 4 | 3
Not completed — Withdrawal by Subject | 4 | 5 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAX-31 Low Dose | VAX-31 Mid Dose | VAX-31 High Dose | PCV20 | Total
Number analyzed (Participants) | 255 | 254 | 253 | 253 | 1015
Age, Continuous [Median (Full Range); unit: years] | 58.0 [50.0 to 84.0] | 58.0 [50.0 to 86.0] | 59.0 [50.0 to 79.0] | 60.0 [50.0 to 82.0] | 59.0 [50.0 to 86.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 160 | 150 | 148 | 609
  Male | 104 | 94 | 103 | 105 | 406
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 44 | 42 | 43 | 172
  Not Hispanic or Latino | 210 | 208 | 209 | 209 | 836
  Unknown or Not Reported | 2 | 2 | 2 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 0 | 0 | 5
  Asian | 3 | 5 | 4 | 3 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 60 | 55 | 51 | 60 | 226
  White | 188 | 191 | 196 | 185 | 760
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 4 | 8
Height (cm) [Median (Inter-Quartile Range); unit: cm] | 167.6 [160.3 to 175.3] | 169.1 [162.6 to 175.3] | 168.0 [162.6 to 175.3] | 167.6 [160.8 to 175.3] | 167.9 [162.5 to 175.3]
Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 82.56 [71.10 to 94.30] | 85.80 [72.00 to 102.15] | 84.00 [71.90 to 99.79] | 83.64 [72.12 to 97.52] | 83.92 [71.90 to 98.80]
Body Mass Index (kg/m^2) [Median (Inter-Quartile Range); unit: kg/m^2] | 28.90 [25.98 to 33.47] | 30.42 [25.58 to 34.42] | 28.82 [25.60 to 33.37] | 29.11 [25.91 to 34.14] | 29.27 [25.78 to 33.91]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Reporting Solicited Local Reactions Within 7 Days After Vaccination (Redness, Swelling, and Pain at Injection Site) in Each Age Group
Description: Solicited local reactions include redness/erythema, swelling/induration, and pain at injection site within 7 days after vaccination in each age group.
Time Frame: 7 days after vaccination
Population: Safety population, defined as all subjects who received study vaccine and provided safety assessment data. Subject safety data were analyzed according to the vaccine as received.
Measure: Number; unit: percentage of participants
Groups:
- VAX-31 Low Dose Overall (Age 50+); VAX-31 Low Dose Age 50-59 Years; VAX-31 Low Dose Age 60+ Years; VAX-31 Low Dose Age 65+ Years: Participants received a single low dose of VAX-31 administered as an intramuscular injection at Day 1.
  1.1 mcg for all serotypes with the exception of serotypes 1, 5, and 22F which is 1.65 mcg.
  31 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-31 will be administered into the deltoid muscle at Day 1
- VAX-31 Mid Dose Overall (Age 50+); VAX-31 Mid Dose Age 50-59 Years; VAX-31 Mid Dose Age 60+ Years; VAX-31 Mid Dose Age 65+ Years: Participants received a single mid dose of VAX-31 administered as an intramuscular injection at Day 1.
  2.2 mcg for all serotypes with the exception of serotypes 1, 5, and 22F which is 3.3 mcg.
  31 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-31 will be administered into the deltoid muscle at Day 1
- VAX-31 High Dose Overall (Age 50+); VAX-31 High Dose Age 50-59 Years; VAX-31 High Dose Age 60+ Years; VAX-31 High Dose Age 65+ Years: Participants received a single high dose of VAX-31 administered as an intramuscular injection at Day 1.
  3.3 mcg for all serotypes with the exception of serotypes 1, 5, and 22F which is 4.4 mcg.
  31 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-31 will be administered into the deltoid muscle at Day 1
- PCV20 Overall (Age 50+); PCV20 Age 50-59 Years; PCV20 Age 60+ Years; PCV20 Age 65+ Years: Participants received a single intramuscular injection of the standard dose of PCV20 at Day 1.
  20 valent pneumococcal conjugate vaccine: 0.5 ml dose of PCV20 will be administered into the deltoid muscle at Day 1
Arm/Group | VAX-31 Low Dose Overall (Age 50+) | VAX-31 Mid Dose Overall (Age 50+) | VAX-31 High Dose Overall (Age 50+) | PCV20 Overall (Age 50+) | VAX-31 Low Dose Age 50-59 Years | VAX-31 Mid Dose Age 50-59 Years | VAX-31 High Dose Age 50-59 Years | PCV20 Age 50-59 Years | VAX-31 Low Dose Age 60+ Years | VAX-31 Mid Dose Age 60+ Years | VAX-31 High Dose Age 60+ Years | PCV20 Age 60+ Years | VAX-31 Low Dose Age 65+ Years | VAX-31 Mid Dose Age 65+ Years | VAX-31 High Dose Age 65+ Years | PCV20 Age 65+ Years
Number analyzed (Participants) | 253 | 254 | 253 | 252 | 145 | 144 | 140 | 116 | 108 | 110 | 113 | 136 | 58 | 59 | 53 | 67
percentage of participants
  Any solicited local AE; Overall, Any Grade | 66.8 | 67.7 | 74.3 | 60.3 | 72.4 | 75.0 | 76.4 | 68.1 | 59.3 | 58.2 | 71.7 | 53.7 | 63.8 | 49.2 | 67.9 | 44.8
  Pain at injection site; Overall, Any Grade | 66.0 | 66.9 | 73.5 | 59.9 | 71.7 | 73.6 | 75.0 | 68.1 | 58.3 | 58.2 | 71.7 | 52.9 | 62.1 | 49.2 | 67.9 | 43.3
  Erythema (redness) at injection site; Overall, Any Grade | 6.3 | 7.5 | 7.1 | 4.4 | 7.6 | 10.4 | 7.1 | 5.2 | 4.6 | 3.6 | 7.1 | 3.7 | 1.7 | 1.7 | 3.8 | 3.0
  Edema (swelling) at injection site; Overall, Any Grade | 5.5 | 7.9 | 7.1 | 3.6 | 6.9 | 7.6 | 7.1 | 5.2 | 3.7 | 8.2 | 7.1 | 2.2 | 1.7 | 5.1 | 5.7 | 0

2. Primary Outcome: Percentage of Subjects Reporting Solicited Systemic Events Within 7 Days After Vaccination (Fever, Headache, Fatigue, Muscle Pain, and Joint Pain) in Each Age Group Vaccination in Each Age Group
Description: Solicited systemic reactions include fever, headache, fatigue, muscle pain, and joint pain.
Time Frame: 7 days after vaccination
Population: Safety population, defined as all subjects who received study vaccine and provided safety assessment data. Subject safety data were analyzed according to the vaccine they received.
Measure: Number; unit: percentage of participants
Arm/Group | VAX-31 Low Dose Overall (Age 50+) | VAX-31 Mid Dose Overall (Age 50+) | VAX-31 High Dose Overall (Age 50+) | PCV20 Overall (Age 50+) | VAX-31 Low Dose Age 50-59 Years | VAX-31 Mid Dose Age 50-59 Years | VAX-31 High Dose Age 50-59 Years | PCV20 Age 50-59 Years | VAX-31 Low Dose Age 60+ Years | VAX-31 Mid Dose Age 60+ Years | VAX-31 High Dose Age 60+ Years | PCV20 Age 60+ Years | VAX-31 Low Dose Age 65+ Years | VAX-31 Mid Dose Age 65+ Years | VAX-31 High Dose Age 65+ Years | PCV20 Age 65+ Years
Number analyzed (Participants) | 253 | 254 | 253 | 252 | 145 | 144 | 140 | 116 | 108 | 110 | 113 | 136 | 58 | 59 | 53 | 67
percentage of participants
  Any solicited systemic AE (any grade) | 58.5 | 61.4 | 68.0 | 57.1 | 64.1 | 65.3 | 71.4 | 59.5 | 50.9 | 56.4 | 63.7 | 55.1 | 50.0 | 54.2 | 60.4 | 55.2
  Fever (any grade) | 1.2 | 1.2 | 1.6 | 0.8 | 1.4 | 1.4 | 2.1 | 0.9 | 0.9 | 0.9 | 0.9 | 0.7 | 1.7 | 1.7 | 0.0 | 0.0
  Fatigue (any grade) | 36.8 | 36.2 | 46.2 | 38.9 | 40.0 | 40.3 | 49.3 | 37.1 | 32.4 | 30.9 | 42.5 | 40.4 | 31.0 | 28.8 | 41.5 | 38.8
  Headache (any grade) | 32.0 | 31.9 | 33.2 | 26.6 | 35.2 | 37.5 | 34.3 | 30.2 | 27.8 | 24.5 | 31.9 | 23.5 | 22.4 | 23.7 | 26.4 | 23.9
  Muscle pain (any grade) | 41.9 | 46.9 | 54.9 | 41.3 | 49.0 | 51.4 | 57.1 | 41.4 | 32.4 | 40.9 | 52.2 | 41.2 | 32.8 | 42.4 | 49.1 | 40.3
  Joint pain (any grade) | 17.4 | 22.0 | 23.3 | 16.7 | 17.9 | 25.7 | 22.9 | 14.7 | 16.7 | 17.3 | 23.9 | 18.4 | 20.7 | 16.9 | 20.8 | 17.9

3. Primary Outcome: Percentage of Subjects Reporting Unsolicited Adverse Event in Each Age Group
Description: Percentage of participants in each age group with adverse events (AEs) whose date of onset occurs after the study vaccine and within the 1 month after vaccination.
Time Frame: 1 month after vaccination
Population: Safety population, defined as all subjects who received study vaccine. Subject safety data were analyzed according to the vaccine they received.
Measure: Number; unit: percentage of participants
Arm/Group | VAX-31 Low Dose Overall (Age 50+) | VAX-31 Mid Dose Overall (Age 50+) | VAX-31 High Dose Overall (Age 50+) | PCV20 Overall (Age 50+) | VAX-31 Low Dose Age 50-59 Years | VAX-31 Mid Dose Age 50-59 Years | VAX-31 High Dose Age 50-59 Years | PCV20 Age 50-59 Years | VAX-31 Low Dose Age 60+ Years | VAX-31 Mid Dose Age 60+ Years | VAX-31 High Dose Age 60+ Years | PCV20 Age 60+ Years | VAX-31 Low Dose Age 65+ Years | VAX-31 Mid Dose Age 65+ Years | VAX-31 High Dose Age 65+ Years | PCV20 Age 65+ Years
Number analyzed (Participants) | 255 | 254 | 253 | 253 | 147 | 144 | 140 | 116 | 108 | 110 | 113 | 137 | 58 | 59 | 53 | 67
percentage of participants | 16.5 | 16.9 | 18.6 | 16.6 | 18.4 | 16.7 | 22.9 | 18.1 | 13.9 | 17.3 | 13.3 | 15.3 | 17.2 | 18.6 | 13.2 | 14.9

4. Primary Outcome: Percentage of Subjects Reporting Serious Adverse Event
Description: Percentage of participants with SAEs.
Time Frame: 6 months after vaccination
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | VAX-31 Low Dose Overall (Age 50+) | VAX-31 Mid Dose Overall (Age 50+) | VAX-31 High Dose Overall (Age 50+) | PCV20 Overall (Age 50+) | VAX-31 Low Dose Age 50-59 Years | VAX-31 Mid Dose Age 50-59 Years | VAX-31 High Dose Age 50-59 Years | PCV20 Age 50-59 Years | VAX-31 Low Dose Age 60+ Years | VAX-31 Mid Dose Age 60+ Years | VAX-31 High Dose Age 60+ Years | PCV20 Age 60+ Years | VAX-31 Low Dose Age 65+ Years | VAX-31 Mid Dose Age 65+ Years | VAX-31 High Dose Age 65+ Years | PCV20 Age 65+ Years
Number analyzed (Participants) | 255 | 254 | 253 | 253 | 147 | 144 | 140 | 116 | 108 | 110 | 113 | 137 | 58 | 59 | 53 | 67
percentage of participants | 0.8 | 1.2 | 2.0 | 1.2 | 1.4 | 0.7 | 2.1 | 0.0 | 0.0 | 1.8 | 1.8 | 2.2 | 0.0 | 1.7 | 3.8 | 3.0

5. Primary Outcome: Percentage of Subjects Reporting New Onset of Chronic Illness
Description: Percentage of participants with NOCIs
Time Frame: 6 months after vaccination
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- VAX-31 Low Dose Age 50+ Years; VAX-31 Low Dose Age 50-59 Years; VAX-31 Low Dose Age 60+ Years; VAX-31 Low Dose Age 65+ Years: Participants received a single low dose of VAX-31 administered as an intramuscular injection at Day 1.
  1.1 mcg for all serotypes with the exception of serotypes 1, 5, and 22F which is 1.65 mcg.
  31 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-31 will be administered into the deltoid muscle at Day 1
- VAX-31 Mid Dose Age 50+ Years; VAX-31 Mid Dose Age 50-59 Years; VAX-31 Mid Dose Age 60+ Years; VAX-31 Mid Dose Age 65+ Years: Participants received a single mid dose of VAX-31 administered as an intramuscular injection at Day 1.
  2.2 mcg for all serotypes with the exception of serotypes 1, 5, and 22F which is 3.3 mcg.
  31 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-31 will be administered into the deltoid muscle at Day 1
- VAX-31 High Dose Age 50+ Years; VAX-31 High Dose Age 50-59 Years; VAX-31 High Dose Age 60+ Years; VAX-31 High Dose Age 65+ Years: Participants received a single high dose of VAX-31 administered as an intramuscular injection at Day 1.
  3.3 mcg for all serotypes with the exception of serotypes 1, 5, and 22F which is 4.4 mcg.
  31 valent pneumococcal conjugate vaccine: 0.5 ml dose of VAX-31 will be administered into the deltoid muscle at Day 1
- PCV20 Age 50+ Years; PCV20 Age 50-59 Years; PCV20 Age 60+ Years; PCV20 Age 65+ Years: Participants received a single intramuscular injection of the standard dose of PCV20 at Day 1.
  20 valent pneumococcal conjugate vaccine: 0.5 ml dose of PCV20 will be administered into the deltoid muscle at Day 1
Arm/Group | VAX-31 Low Dose Age 50+ Years | VAX-31 Mid Dose Age 50+ Years | VAX-31 High Dose Age 50+ Years | PCV20 Age 50+ Years | VAX-31 Low Dose Age 50-59 Years | VAX-31 Mid Dose Age 50-59 Years | VAX-31 High Dose Age 50-59 Years | PCV20 Age 50-59 Years | VAX-31 Low Dose Age 60+ Years | VAX-31 Mid Dose Age 60+ Years | VAX-31 High Dose Age 60+ Years | PCV20 Age 60+ Years | VAX-31 Low Dose Age 65+ Years | VAX-31 Mid Dose Age 65+ Years | VAX-31 High Dose Age 65+ Years | PCV20 Age 65+ Years
Number analyzed (Participants) | 255 | 254 | 253 | 253 | 147 | 144 | 140 | 116 | 108 | 110 | 113 | 137 | 58 | 59 | 53 | 67
percentage of participants | 0.8 | 2.4 | 2.0 | 2.0 | 0.0 | 1.4 | 2.1 | 0.9 | 1.9 | 3.6 | 1.8 | 2.9 | 3.4 | 3.4 | 1.9 | 1.5

6. Primary Outcome: Percentage of Subjects Reporting Medically Attended Adverse Event
Description: Percentage of participants with MAAEs.
Time Frame: 6 months after vaccination
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | VAX-31 Low Dose Overall (Age 50+) | VAX-31 Mid Dose Overall (Age 50+) | VAX-31 High Dose Overall (Age 50+) | PCV20 Overall (Age 50+) | VAX-31 Low Dose Age 50-59 Years | VAX-31 Mid Dose Age 50-59 Years | VAX-31 High Dose Age 50-59 Years | PCV20 Age 50-59 Years | VAX-31 Low Dose Age 60+ Years | VAX-31 Mid Dose Age 60+ Years | VAX-31 High Dose Age 60+ Years | PCV20 Age 60+ Years | VAX-31 Low Dose Age 65+ Years | VAX-31 Mid Dose Age 65+ Years | VAX-31 High Dose Age 65+ Years | PCV20 Age 65+ Years
Number analyzed (Participants) | 255 | 254 | 253 | 253 | 147 | 144 | 140 | 116 | 108 | 110 | 113 | 137 | 58 | 59 | 53 | 67
percentage of participants | 17.6 | 16.5 | 13.8 | 12.3 | 17.0 | 18.1 | 15.0 | 13.8 | 18.5 | 14.5 | 12.4 | 10.9 | 22.4 | 15.3 | 9.4 | 11.9

7. Secondary Outcome: Percentage of Subjects With Adverse Events Due to Clinically Significant Laboratory Values
Description: Laboratory values that resulted in treatment and reporting as adverse events 1 month following vaccination.
Time Frame: 1 month after vaccination
Population: Safety population, including all subjects who received study vaccine and provided safety assessment data. Subject safety data were analyzed according to the vaccine they received.
Measure: Count of Participants; unit: Participants
Arm/Group | VAX-31 Low Dose | VAX-31 Mid Dose | VAX-31 High Dose | PCV20
Number analyzed (Participants) | 255 | 254 | 253 | 253
Participants
  Hemoglobin (low) | 0 | 0 | 1 | 0
  Platelets (low) | 0 | 1 | 0 | 0
  Platelets (high) | 0 | 0 | 1 | 0
  Leukocytes (low) | 0 | 0 | 0 | 1
  Leukocytes (high) | 0 | 0 | 0 | 0
  Alanine aminotransferase (high) | 1 | 0 | 1 | 1
  Aspartate aminotransferase (high) | 1 | 0 | 1 | 0
  Cholesterol (high) | 0 | 1 | 0 | 0
  Creatinine (high) | 0 | 1 | 0 | 0
  Gamma glutamyl transferase (high) | 0 | 0 | 1 | 1
  Glucose (low) | 1 | 0 | 0 | 0
  Glucose (high) | 1 | 0 | 0 | 1
  Potassium (low) | 0 | 1 | 0 | 0
  Potassium (high) | 1 | 0 | 0 | 0
  Sodium (low) | 0 | 0 | 1 | 0
  Triglycerides (high) | 1 | 0 | 1 | 0
  Urine glucose | 0 | 1 | 0 | 0
  Urine hemoglobin | 1 | 2 | 1 | 2
  Eosinophils | 0 | 0 | 0 | 0
  Neutrophils | 0 | 0 | 0 | 0
  Alkaline phosphatase | 0 | 0 | 0 | 0
  Albumin | 0 | 0 | 0 | 0
  Bicarbonate | 0 | 0 | 0 | 0
  Bilirubin | 0 | 0 | 0 | 0
  Direct bilirubin | 0 | 0 | 0 | 0
  Calcium | 0 | 0 | 0 | 0
  Chloride | 0 | 0 | 0 | 0
  Lactate dehydrogenase | 0 | 0 | 0 | 0
  Phosphate | 0 | 0 | 0 | 0
  Protein | 0 | 0 | 0 | 0
  Urate | 0 | 0 | 0 | 0
  Urea nitrogen | 0 | 0 | 0 | 0
  Ketones | 0 | 0 | 0 | 0
  Leukocyte esterase | 0 | 0 | 0 | 0
  Urine bilirubin | 0 | 0 | 0 | 0
  Urine protein | 0 | 0 | 0 | 0
  Nitrite | 0 | 0 | 0 | 0
  Urobilinogen | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants With a Shift From Normal at Baseline to Abnormal at Post-vaccination in Safety Laboratory Parameters (Hematology, Clinical Chemistry, Urinalysis)
Description: Shifts from Normal at Baseline to Abnormal on Month 1 (30 days after vaccination) in Hematology, Clinical Chemistry and Urinalysis Parameters Occurring in Subjects Aged 50+ Years.
Time Frame: 1 month after vaccination
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | VAX-31 Low Dose | VAX-31 Mid Dose | VAX-31 High Dose | PCV20
Number analyzed (Participants) | 255 | 254 | 253 | 253
percentage of participants
  Eosinophils (10^9/L) | 1.6 | 1.2 | 1.6 | 0.0
  Hemoglobin (g/L) | 2.8 | 1.2 | 4.0 | 1.2
  Neutrophils (10^9/L) | 5.1 | 4.7 | 5.1 | 2.0
  Platelets (10^9/L) | 1.2 | 2.0 | 1.2 | 0.0
  Leukocytes (10^9/L) | 6.3 | 4.7 | 4.7 | 4.3
  Albumin (g/L) | 0.0 | 0.0 | 0.0 | 0.4
  Alkaline phosphatase (U/L) | 2.4 | 1.6 | 1.6 | 0.8
  Alanine aminotransferase (U/L) | 2.4 | 4.3 | 2.0 | 2.0
  Aspartate aminotransferase (U/L) | 2.0 | 2.0 | 0.4 | 2.4
  Bicarbonate (mmol/L) | 1.2 | 2.0 | 2.0 | 3.2
  Direct bilirubin (umol/L) | 0.8 | 0.0 | 0.4 | 0.0
  Bilirubin (umol/L) | 1.2 | 0.8 | 0.4 | 0.0
  Calcium (mmol/L) | 6.7 | 5.9 | 7.1 | 5.9
  Cholesterol (mmol/L) | 5.1 | 6.7 | 4.0 | 5.5
  Chloride (mmol/L) | 3.1 | 3.9 | 6.3 | 2.4
  Creatinine (umol/L) | 9.0 | 5.5 | 9.5 | 10.3
  Gamma glutamyl transferase (U/L) | 1.6 | 2.0 | 1.2 | 2.0
  Glucose (mmol/L) | 18.0 | 21.3 | 21.0 | 24.1
  Potassium (mmol/L) | 3.5 | 2.8 | 2.8 | 2.8
  Lactate dehydrogenase (U/L) | 0.4 | 0.4 | 0.0 | 0.4
  Phosphate (mmol/L) | 5.9 | 3.2 | 5.2 | 4.8
  Protein (g/L) | 1.2 | 1.6 | 1.2 | 2.8
  Sodium (mmol/L) | 3.9 | 3.1 | 4.0 | 2.8
  Triglycerides (mmol/L) | 6.7 | 9.1 | 7.5 | 8.7
  Urate (umol/L) | 7.1 | 7.9 | 6.3 | 6.7
  Urea nitrogen (mmol/L) | 7.5 | 5.1 | 7.5 | 8.7
  Ketones | 1.6 | 0.8 | 0.0 | 1.2
  Leukocyte esterase | 6.5 | 7.1 | 7.8 | 8.3
  Urine bilirubin | 1.2 | 2.4 | 2.0 | 1.6
  Urine glucose | 0.8 | 0.8 | 1.3 | 0.8
  Urine hemoglobin | 1.2 | 2.4 | 2.4 | 2.5
  Urine protein | 1.2 | 2.0 | 2.0 | 3.7
  Nitrite | 0.4 | 1.2 | 2.8 | 0.8
  Urobilinogen | 0.0 | 0.4 | 0.0 | 0.0

9. Secondary Outcome: 31 VAX-31 Pneumococcal Serotype-specific OPA Geometric Mean Titer
Description: Antibody geometric mean titers as measured by OPA for the 31 pneumococcal serotypes in VAX-31.
Time Frame: 1 month after vaccination
Population: Immunogenicity Evaluable Population included all subjects 50+ years who received study vaccine, with no major protocol deviation impacting immunogenicity assessment, no prohibited medication or vaccine, and provided evaluable serum sample results for baseline and Month 1 within required time frames. Data were analyzed according to vaccine received.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | VAX-31 Low Dose | VAX-31 Mid Dose | VAX-31 High Dose | PCV20
Number analyzed (Participants) | 247 | 245 | 244 | 247
mcg/mL
  1: number analyzed (Participants) | 247 | 244 | 244 | 244
  1 | 412.94 [346.34 to 492.35] | 474.22 [397.08 to 566.36] | 509.76 [426.79 to 608.85] | 410.32 [343.55 to 490.06]
  2: number analyzed (Participants) | 247 | 244 | 244 | 244
  2 | 1984.89 [1687.63 to 2334.51] | 2158.32 [1830.96 to 2544.21] | 2376.00 [2016.93 to 2798.99] | 160.47 [136.23 to 189.01]
  3: number analyzed (Participants) | 240 | 241 | 240 | 241
  3 | 247.34 [215.11 to 284.39] | 301.19 [261.87 to 346.41] | 369.12 [320.89 to 424.61] | 351.45 [305.59 to 404.18]
  4: number analyzed (Participants) | 247 | 245 | 244 | 246
  4 | 1909.83 [1697.83 to 2148.29] | 1923.46 [1708.37 to 2165.64] | 2204.29 [1957.32 to 2482.43] | 1909.84 [1696.64 to 2149.82]
  5: number analyzed (Participants) | 247 | 245 | 244 | 246
  5 | 453.32 [366.56 to 560.62] | 553.68 [446.96 to 685.89] | 643.83 [519.50 to 797.91] | 518.71 [418.91 to 642.29]
  6A: number analyzed (Participants) | 247 | 243 | 243 | 244
  6A | 3017.66 [2421.39 to 3760.77] | 3649.18 [2920.00 to 4560.43] | 5476.69 [4383.39 to 6842.69] | 5039.25 [4034.70 to 6293.90]
  6B: number analyzed (Participants) | 245 | 240 | 238 | 243
  6B | 3114.80 [2534.60 to 3827.81] | 3430.49 [2784.90 to 4225.76] | 4778.40 [3874.70 to 5892.86] | 4032.19 [3277.67 to 4960.39]
  7C: number analyzed (Participants) | 247 | 245 | 243 | 233
  7C | 5333.37 [4722.15 to 6023.70] | 5642.80 [4991.20 to 6379.48] | 6230.76 [5507.58 to 7048.89] | 656.15 [578.74 to 743.90]
  7F: number analyzed (Participants) | 240 | 238 | 240 | 241
  7F | 4889.66 [4224.12 to 5660.06] | 5647.05 [4857.85 to 6540.22] | 6584.45 [5686.59 to 7624.08] | 4990.65 [4311.96 to 5776.16]
  8: number analyzed (Participants) | 245 | 240 | 235 | 244
  8 | 1614.83 [1399.07 to 1863.87] | 1943.14 [1680.15 to 2247.28] | 2329.26 [2010.27 to 2698.88] | 2077.75 [1798.13 to 2400.84]
  9N: number analyzed (Participants) | 246 | 245 | 243 | 239
  9N | 6245.38 [5374.40 to 7257.52] | 7075.75 [6082.90 to 8230.66] | 7924.85 [6808.85 to 9223.76] | 1484.59 [1274.23 to 1729.67]
  9V: number analyzed (Participants) | 245 | 245 | 244 | 246
  9V | 4709.89 [4015.67 to 5524.13] | 5572.21 [4748.00 to 6539.50] | 5353.40 [4560.06 to 6284.77] | 3700.19 [3153.92 to 4341.07]
  10A: number analyzed (Participants) | 246 | 244 | 244 | 247
  10A | 2718.18 [2272.32 to 3251.53] | 4553.86 [3800.58 to 5456.44] | 4715.10 [3936.02 to 5648.37] | 4849.53 [4052.41 to 5803.44]
  11A: number analyzed (Participants) | 244 | 242 | 243 | 240
  11A | 1130.91 [1061.75 to 1204.58] | 1101.72 [1033.84 to 1174.07] | 1147.21 [1076.37 to 1222.72] | 946.05 [887.55 to 1008.41]
  12F: number analyzed (Participants) | 244 | 240 | 238 | 242
  12F | 1199.57 [968.68 to 1485.49] | 1389.71 [1119.73 to 1724.78] | 1658.63 [1335.19 to 2060.42] | 1382.15 [1115.80 to 1712.08]
  14: number analyzed (Participants) | 245 | 243 | 242 | 246
  14 | 3574.38 [3048.13 to 4191.50] | 4000.68 [3404.71 to 4700.99] | 4657.38 [3965.48 to 5469.99] | 4306.60 [3670.73 to 5052.62]
  15A: number analyzed (Participants) | 242 | 243 | 236 | 238
  15A | 8705.55 [7402.46 to 10238.03] | 9982.41 [8488.71 to 11738.94] | 10153.26 [8613.07 to 11968.86] | 2696.64 [2290.66 to 3174.58]
  15B: number analyzed (Participants) | 233 | 229 | 231 | 232
  15B | 2891.81 [2423.77 to 3450.24] | 3548.99 [2969.28 to 4241.87] | 3877.44 [3243.71 to 4634.98] | 2568.68 [2149.28 to 3069.93]
  16F: number analyzed (Participants) | 247 | 245 | 244 | 244
  16F | 7931.81 [6996.40 to 8992.27] | 9980.42 [8794.73 to 11325.96] | 11055.25 [9739.33 to 12548.96] | 2130.17 [1876.88 to 2417.65]
  17F: number analyzed (Participants) | 247 | 244 | 242 | 235
  17F | 2146.39 [1904.03 to 2419.61] | 2112.12 [1871.11 to 2384.19] | 2160.76 [1913.48 to 2439.99] | 405.86 [358.82 to 459.08]
  18C: number analyzed (Participants) | 242 | 243 | 244 | 244
  18C | 1928.40 [1599.06 to 2325.57] | 2302.99 [1910.36 to 2776.31] | 2640.00 [2190.27 to 3182.06] | 1845.17 [1531.20 to 2223.52]
  19A | 4199.53 [3606.89 to 4889.55] | 4726.99 [4055.05 to 5510.27] | 5032.82 [4316.05 to 5868.63] | 4271.98 [3666.77 to 4977.07]
  19F | 1754.37 [1541.08 to 1997.18] | 1817.82 [1595.18 to 2071.52] | 2185.14 [1917.00 to 2490.78] | 1321.85 [1160.51 to 1505.61]
  20B: number analyzed (Participants) | 244 | 241 | 244 | 240
  20B | 9756.59 [8193.85 to 11617.39] | 10664.95 [8936.58 to 12727.60] | 9988.69 [8381.50 to 11904.07] | 427.17 [358.03 to 509.66]
  22F: number analyzed (Participants) | 247 | 245 | 243 | 247
  22F | 7196.50 [6125.39 to 8454.92] | 8843.18 [7517.43 to 10402.73] | 8633.65 [7333.92 to 10163.72] | 9989.08 [8496.59 to 11743.74]
  23A: number analyzed (Participants) | 243 | 241 | 240 | 223
  23A | 2778.60 [2235.23 to 3454.05] | 2929.12 [2354.16 to 3644.51] | 3253.49 [2612.93 to 4051.07] | 175.01 [139.54 to 219.49]
  23B: number analyzed (Participants) | 237 | 236 | 234 | 229
  23B | 1919.13 [1555.79 to 2367.32] | 1855.53 [1501.21 to 2293.47] | 2010.19 [1625.78 to 2485.48] | 248.33 [200.25 to 307.96]
  23F: number analyzed (Participants) | 245 | 244 | 244 | 247
  23F | 1829.26 [1475.00 to 2268.62] | 2128.26 [1714.84 to 2641.34] | 2491.49 [2007.55 to 3092.09] | 1433.09 [1156.18 to 1776.33]
  31: number analyzed (Participants) | 247 | 245 | 244 | 237
  31 | 7199.08 [5973.44 to 8676.19] | 7821.34 [6480.26 to 9439.94] | 8605.44 [7127.04 to 10390.50] | 623.66 [515.16 to 755.00]
  33F: number analyzed (Participants) | 231 | 226 | 233 | 234
  33F | 10686.74 [9102.59 to 12546.58] | 12553.75 [10684.65 to 14749.82] | 12763.17 [10869.89 to 14986.22] | 10332.19 [8815.38 to 12109.97]
  35B: number analyzed (Participants) | 247 | 245 | 244 | 242
  35B | 9264.48 [8193.76 to 10475.12] | 9913.10 [8758.88 to 11219.41] | 10659.18 [9415.66 to 12066.95] | 2845.55 [2511.80 to 3223.64]

10. Secondary Outcome: 31 VAX-31 Pneumococcal Serotype-specific IgG Geometric Mean Concentration
Description: Antibody geometric mean concentrations as measured by IgG for the 31 pneumococcal serotypes in VAX-31.
Time Frame: 1 month after vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | VAX-31 Low Dose | VAX-31 Mid Dose | VAX-31 High Dose | PCV20
Number analyzed (Participants) | 247 | 245 | 244 | 247
mcg/mL
  1 | 5.56 [4.78 to 6.48] | 5.55 [4.76 to 6.48] | 6.40 [5.49 to 7.46] | 4.32 [3.71 to 5.04]
  2: number analyzed (Participants) | 247 | 245 | 244 | 244
  2 | 12.64 [10.60 to 15.08] | 14.78 [12.37 to 17.66] | 15.04 [12.59 to 17.97] | 0.93 [0.78 to 1.11]
  3: number analyzed (Participants) | 247 | 245 | 243 | 247
  3 | 0.47 [0.40 to 0.55] | 0.53 [0.45 to 0.61] | 0.61 [0.52 to 0.71] | 0.60 [0.52 to 0.70]
  4 | 1.22 [1.02 to 1.46] | 1.56 [1.30 to 1.86] | 1.73 [1.44 to 2.06] | 1.50 [1.26 to 1.79]
  5 | 2.38 [2.01 to 2.83] | 2.82 [2.38 to 3.35] | 2.80 [2.36 to 3.33] | 2.47 [2.08 to 2.93]
  6A: number analyzed (Participants) | 246 | 243 | 244 | 244
  6A | 2.97 [2.42 to 3.66] | 3.15 [2.56 to 3.89] | 4.28 [3.48 to 5.27] | 3.14 [2.55 to 3.87]
  6B: number analyzed (Participants) | 246 | 244 | 244 | 243
  6B | 3.26 [2.58 to 4.13] | 3.88 [3.06 to 4.92] | 5.01 [3.95 to 6.35] | 3.08 [2.43 to 3.91]
  7C: number analyzed (Participants) | 247 | 245 | 243 | 244
  7C | 11.96 [9.47 to 15.09] | 14.02 [11.09 to 17.73] | 13.71 [10.83 to 17.36] | 0.56 [0.44 to 0.71]
  7F: number analyzed (Participants) | 246 | 245 | 244 | 245
  7F | 5.81 [4.97 to 6.80] | 6.59 [5.63 to 7.72] | 7.10 [6.06 to 8.32] | 5.14 [4.39 to 6.01]
  8: number analyzed (Participants) | 247 | 245 | 243 | 247
  8 | 6.13 [5.24 to 7.16] | 7.44 [6.36 to 8.70] | 9.69 [8.27 to 11.34] | 6.99 [5.97 to 8.17]
  9N: number analyzed (Participants) | 246 | 245 | 244 | 245
  9N | 6.52 [5.49 to 7.73] | 6.60 [5.56 to 7.84] | 7.92 [6.67 to 9.41] | 1.00 [0.84 to 1.19]
  9V: number analyzed (Participants) | 243 | 244 | 240 | 246
  9V | 3.77 [3.12 to 4.55] | 4.31 [3.57 to 5.20] | 3.78 [3.12 to 4.57] | 2.63 [2.18 to 3.17]
  10A: number analyzed (Participants) | 246 | 245 | 242 | 247
  10A | 6.67 [5.27 to 8.43] | 7.55 [5.96 to 9.56] | 8.21 [6.47 to 10.40] | 10.82 [8.55 to 13.69]
  11A: number analyzed (Participants) | 247 | 245 | 244 | 246
  11A | 4.78 [4.00 to 5.71] | 5.70 [4.76 to 6.82] | 5.37 [4.49 to 6.42] | 3.75 [3.13 to 4.48]
  12F | 1.52 [1.24 to 1.86] | 1.96 [1.60 to 2.40] | 1.70 [1.39 to 2.08] | 1.38 [1.13 to 1.68]
  14 | 7.41 [6.02 to 9.12] | 10.33 [8.38 to 12.74] | 11.58 [9.38 to 14.28] | 9.15 [7.42 to 11.27]
  15A: number analyzed (Participants) | 247 | 245 | 243 | 247
  15A | 20.93 [17.27 to 25.38] | 26.40 [21.75 to 32.06] | 25.91 [21.32 to 31.50] | 4.22 [3.48 to 5.12]
  15B | 12.34 [10.04 to 15.16] | 4.06 [3.45 to 4.79] | 18.25 [14.82 to 22.46] | 13.17 [10.71 to 16.19]
  16F: number analyzed (Participants) | 247 | 245 | 243 | 247
  16F | 3.03 [2.57 to 3.57] | 4.06 [3.45 to 4.79] | 3.82 [3.24 to 4.51] | 0.95 [0.81 to 1.12]
  17F: number analyzed (Participants) | 247 | 245 | 244 | 246
  17F | 9.54 [8.08 to 11.27] | 11.05 [9.35 to 13.06] | 12.67 [10.72 to 14.99] | 0.56 [0.47 to 0.66]
  18C | 7.15 [5.91 to 8.67] | 8.34 [6.87 to 10.11] | 8.31 [6.85 to 10.09] | 6.62 [5.46 to 8.03]
  19A: number analyzed (Participants) | 246 | 245 | 244 | 247
  19A | 8.08 [6.64 to 9.83] | 11.00 [9.03 to 13.39] | 11.83 [9.71 to 14.41] | 8.53 [7.01 to 10.38]
  19F: number analyzed (Participants) | 246 | 245 | 243 | 245
  19F | 5.94 [4.82 to 7.34] | 6.94 [5.62 to 8.58] | 8.91 [7.20 to 11.02] | 4.37 [3.54 to 5.40]
  20B | 16.33 [13.89 to 19.19] | 20.44 [17.37 to 24.05] | 20.24 [17.20 to 23.83] | 3.91 [3.33 to 4.60]
  22F: number analyzed (Participants) | 247 | 245 | 243 | 246
  22F | 3.45 [2.93 to 4.06] | 4.05 [3.43 to 4.77] | 4.60 [3.90 to 5.43] | 4.37 [3.71 to 5.16]
  23A | 3.05 [2.43 to 3.84] | 3.23 [2.57 to 4.07] | 4.01 [3.18 to 5.05] | 0.52 [0.42 to 0.66]
  23B | 23.14 [19.65 to 27.27] | 25.41 [21.54 to 29.97] | 28.61 [24.25 to 33.76] | 11.27 [9.56 to 13.29]
  23F: number analyzed (Participants) | 247 | 245 | 243 | 246
  23F | 4.58 [3.79 to 5.53] | 5.51 [4.56 to 6.66] | 6.45 [5.33 to 7.80] | 4.60 [3.81 to 5.56]
  31: number analyzed (Participants) | 247 | 245 | 243 | 247
  31 | 6.84 [5.64 to 8.31] | 10.46 [8.61 to 12.72] | 11.92 [9.80 to 14.50] | 0.44 [0.36 to 0.53]
  33F | 13.10 [11.12 to 15.43] | 14.21 [12.05 to 16.76] | 15.88 [13.46 to 18.73] | 12.24 [10.39 to 14.43]
  35B: number analyzed (Participants) | 247 | 245 | 243 | 246
  35B | 25.39 [21.52 to 29.96] | 31.05 [26.28 to 36.68] | 36.39 [30.77 to 43.03] | 3.05 [2.58 to 3.60]

ADVERSE EVENTS:
Time Frame: 6 months
Description: All subjects had safety labs analyzed at Baseline and 1 month post-vaccination. Solicited AEs were collected for 7 days and unsolicited AEs for 1 month post-vaccination. SAEs, new onset of chronic illness and medically attended adverse events were collected for 6 months post-vaccination. Subject safety data were analyzed according to the vaccine regimen received.
Arm/Group | VAX-31 Low Dose Overall (Age 50+) | VAX-31 Mid Dose Overall (Age 50+) | VAX-31 High Dose Overall (Age 50+) | PCV20 Overall (Age 50+)
All-Cause Mortality (participants affected / at risk) | 0/255 | 0/254 | 0/253 | 0/253
Serious Adverse Events (participants affected / at risk) | 2/255 | 3/254 | 5/253 | 3/253
Other Adverse Events (participants affected / at risk) | 189/255 | 196/254 | 209/253 | 178/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAX-31 Low Dose Overall (Age 50+) (N=255) | VAX-31 Mid Dose Overall (Age 50+) (N=254) | VAX-31 High Dose Overall (Age 50+) (N=253) | PCV20 Overall (Age 50+) (N=253)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | VAX-31 Low Dose Overall (Age 50+) (N=255) | VAX-31 Mid Dose Overall (Age 50+) (N=254) | VAX-31 High Dose Overall (Age 50+) (N=253) | PCV20 Overall (Age 50+) (N=253)
Pain at injection site (Skin and subcutaneous tissue disorders) | 167 (167) | 170 (170) | 186 (186) | 151/252 (151)
Erythema (Skin and subcutaneous tissue disorders) | 16 (16) | 19 (19) | 18 (18) | 11/252 (11)
Edema (Skin and subcutaneous tissue disorders) | 14 (14) | 20 (20) | 18 (18) | 9/252 (9)
Fever (General disorders) | 3 (3) | 3 (3) | 4 (4) | 2/252 (2)
Headache (General disorders) | 81 (81) | 81 (81) | 84 (84) | 67/252 (67)
Tiredness (General disorders) | 93 (93) | 92 (92) | 117 (117) | 98/252 (98)
Muscle pain (Musculoskeletal and connective tissue disorders) | 106 (106) | 119 (119) | 139 (139) | 104/252 (104)
Joint pain (Musculoskeletal and connective tissue disorders) | 44 (44) | 56 (56) | 59 (59) | 42/252 (42)
Injection site pruritis (General disorders) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Some limitations of this clinical study include the lack of a group, such as 3.3 mcg or 4.4 mcg, for all serotypes, aimed at understanding whether the dose response of polysaccharide can overcome carrier suppression. The relatively low ethnic diversity of participants is also a limitation, which will be addressed in larger phase 3 clinical trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall review within the ninety (90) day period. Upon receiving any notification from Sponsor requesting deletion of Confidential Information, correction of inaccuracies, or a delay in publication to allow the filing of patent application, Institution or Investigator shall take the requested action of Sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT06151288/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT06151288/SAP_001.pdf